CLINICAL TRIAL: NCT06051669
Title: Comparison of iLivTouch and FibroScan for the Assessment of Liver Fibrosis and Steatosis in Adult Patients in the US: A Multicenter, Cross-sectional, and Prospective Study
Brief Title: Comparison of iLivTouch and FibroScan for the Assessment of Liver Fibrosis and Steatosis in Adult Patients in the US
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: New Discovery LLC (Industry)
Collaborators: NYU Langone Health (Other); Stanford University (Other); Rush University (Other); Baylor University (Other); Wuxi Hisky Medical Technology Co Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ILT-US-2023-01
Record Dates: First submitted 2023-09-01; First posted 2023-09-25 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Liver Fibrosis; Fatty Liver
MeSH Terms: conditions — Liver Cirrhosis; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- iLivTouch then FibroScan: Subjects in the Group "iLivTouch then FibroScan" will be measured using iLivTouch first and then FibroScan based on the randomization result.
  Interventions: Device: iLivTouch; Device: FibroScan
- FibroScan then iLivTouch: Subjects in the Group "FibroScan then iLivTouch" will be measured using FibroScan first and then iLivTouch based on the randomization result.
  Interventions: Device: iLivTouch; Device: FibroScan

INTERVENTIONS:
Device: iLivTouch — The examination with iLivTouch will be performed in each subject following the sequence determined by the randomization results.
Device: FibroScan — The examination with FibroScan will be performed in each subject following the sequence determined by the randomization results.

SUMMARY:
This is a multi-center, cross-sectional, and prospective study that will recruit patients from multiple hospitals or outpatient clinics in the USA to the comparison of iLivTouch and FibroScan for the assessment of liver fibrosis and steatosis in adult patients.

DETAILED DESCRIPTION:
Clinical phase: Phase IV investigator-initiated study Study centers planned: Approximately 4 centers in different regions of the USA

Objectives:

1. Primary Objectives To evaluate the consistency of Liver Stiffness Measurement (LSM) and Ultrasound/Controlled Attenuation Parameters (UAP/CAP) between iLivTouch-FT9000 and FibroScan 530 devices.
2. Secondary Objectives

   1. To compare the operational features of the two devices, reflected in the success rate of examination and number of effective examinations.
   2. To compare LSM obtained from each device with liver stiffness estimated by APRI, FIB-4, and SAFE scores.
   3. The number of adverse events, serious events, and percentage of subjects with events will be calculated for AE, SAE, AE of special interest, and AE leading to study withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* a. Adults aged above 18 years old who have at least one indication for TE examination determined by the physicians;
* b. Patients who have test results for platelet count, ALT, AST, globulin, HBA1c, and total bilirubin (TBIL) levels within 60 days;
* c. Patients who are willing to participate in the clinical study and can sign ICF.

Exclusion Criteria:

* a. Excessive drinking history within 90 days: For women-140 grams of alcohol per week or more; For men-210 grams of alcohol per week or more;
* b. Patients with alanine aminotransferase (ALT) or aspartate aminotransferase AST >100 U/ml (or 2.5 × upper limit of normal (ULN) and/or total bilirubin (TBIL) > 1.8 mg/d (or >1.5 × ULN =1.2 mg/d);
* c. Patients with a history or current evidence of decompensated liver cirrhosis;
* d. Patients with various space-occupying tumors and cysts in the right liver;
* e. Patients with other serious systemically diseases or a history of malignant tumors;
* f. Patients with ascites;
* g. Patients with a non-healing wound on the right upper abdomen at this moment;
* h. Patients with intracavitary implantation of instruments;
* i. Pregnant women (urine pregnancy test should be performed for all women with child-bearing potential during screening);
* j. Any history of organ transplantation and existing functional grafts (except corneal or hair transplantation);
* k. Lack of or limited legal capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adults aged above 18 years old who have at least one indication for TE examination determined by the physicians
Study Population: The following conditions are considered as patient withdrawal from the current study:
  * Patient withdrawal of informed consent at any time during the study;
  * The lack of adherence to the protocol to complete the tests by two devices.
Sampling Method: Non-Probability Sample
Enrollment: 418 (Estimated)
Dates: Start 2023-09-24 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Liver Stiffness Measurement (LSM) value from iLivTouch and FibroScan detection | 6 months
  Spearman correlation coefficients and 95% confidence interval will be calculated to analyze the correlation of the measurements (LSM) between iLivTouch-FT9000 and FibroScan 530 devices.
Ultrasound/Controlled Attenuation Parameters (UAP/CAP) from iLivTouch and FibroScan detection | 6 months
  Spearman correlation coefficients and 95% confidence interval will be calculated to analyze the correlation of the measurements (UAP/CAP) between iLivTouch-FT9000 and FibroScan 530 devices.

SECONDARY OUTCOMES:
To compare the success rate of the iLivTouch and FibroScan | 6 months
  The success rate of examination will be obtained from the percentage of patients who are successful in the test.
To compare the number of effective examinations of iLivTouch and FibroScan | 6 months
  The number of effective examinations will be obtained from the number of attempts to obtain the effective results.
Liver stiffness measurement (LSM) and AST to Platelet Ratio Index (APRI) | 6 months
  To compare LSM obtained from each device with liver stiffness estimated by APRI.
  Two liver fibrosis detection results based on LSM and APRI will be compared. The higher values mean more serious fibrosis.
Liver stiffness measurement (LSM) and Fibrosis-4 (FIB-4) | 6 months
  Two liver fibrosis detection results based on LSM and FIB-4 will be compared. FIB-4 refers to Age (years), AST Level (U/L), Platelet Count (10^9/L), ALT (U/L), with higher values mean more serious fibrosis.
Liver stiffness measurement (LSM) and Steatosis-associated Fibrosis Estimator (SAFE) scores | 6 months
  Two liver fibrosis detection results based on LSM and SAFE scores will be compared. The higher values mean more serious fibrosis.
Adverse events, serious events | 6 months
  The number of adverse events, serious events, and percentage of subjects with events will be calculated for AE, SAE, AE of special interest, and AE leading to study withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Calvin Q. Pan, Study Chair — New York University Langone Health
Locations (4):
- United States (4):
  - Stanford University, Redwood City, California
  - Rush University, Chicago, Illinois
  - NYU Langone, New York, New York
  - Baylor University, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided